CLINICAL TRIAL: NCT02247388
Title: Automated Bilingual Computerized Alcohol Screen and Intervention in Latinos
Brief Title: Automated Bilingual Computerized Alcohol Screening and Intervention in Latinos (AB-CASI)
Acronym: AB-CASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1211011052; R01AA022083-01A1 (NIH)
Record Dates: First submitted 2014-09-16; First posted 2014-09-25 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Dependence; Alcoholism; AB-CASI; Emergency Department
MeSH Terms: conditions — Alcoholism; Emergencies | interventions — Ethanol; Mass Screening

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AB-CASI (Experimental): Automated Bilingual Computerized Alcohol Screening and Brief Negotiated Interview(BNI) Intervention
  Interventions: Behavioral: Computerized Alcohol Screening; Behavioral: Brief Negotiated Interview
- Standard Care (No Intervention): Standard Care

INTERVENTIONS:
Behavioral: Computerized Alcohol Screening — iPad based automated alcohol screening
  Arms: AB-CASI
Behavioral: Brief Negotiated Interview — iPad based automated brief negotiated interview (BNI)
  Other Names: BNI
  Arms: AB-CASI

SUMMARY:
To study the efficacy of AB-CASI against standard of care in a randomized controlled trial in the Emergency Department.

DETAILED DESCRIPTION:
The research team will rigorously test the efficacy of AB-CASI, against a standard condition (SC) in a first-of-a-kind ED randomized controlled trial. Studying an urban adult (≥ 18 y/o) Latino ED population, the objectives are to demonstrate the superiority of AB-CASI compared to SC in: 1) reduction of alcohol consumption (Aims 1), 2) reduction of negative health behaviors and consequences (Aim 2), and 3) increasing 30-day treatment engagement (Aim 3). The investigators will also explore variation of the AB-CASI intervention on alcohol consumption, alcohol-related negative health behaviors and consequences, and 30-day treatment engagement by Latino subpopulations (Puerto-Rican, Mexican-American, Cuban-American, South/Central American) as well as other potential modifiers (age, birthplace, gender, preferred language, reason for ED visit, and smoking status). English and Spanish speaking Latino adults presenting to the Bridgeport Hospital ED will be screened using the study inclusion and exclusion criteria.

In March 2020, the primary and secondary outcomes were corrected to reflect the protocol as it was written initially. The citations section of this study registration also includes the citation for the published protocol manuscript.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish speaking adult
* ≥ 18 y/o
* Latino patients who present to the Bridgeport Hospital's ED
* Drink over the NIAAA low-risk limits.

Exclusion Criteria:

* Primary language other than English or Spanish
* Current enrollment in an alcohol or substance abuse treatment program
* Current ED visit for acute psychosis
* Condition that precludes interview or AB-CASI use i.e., life threatening injury/illness
* In police custody
* Inability to provide two contact numbers for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2014-10; Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Self Reported Binge Drinking Episodes | 12 months
  Self reported number of binge drinking episodes over the previous 28 days assessed using the 28 day timeline follow back at 12 months.
  This outcome was corrected 3/2020 to accurately reflect the time frame from the original protocol.

SECONDARY OUTCOMES:
Mean Number of Weekly Drinks | 12 months post enrollment
  Self reported mean number of weekly drinks as measured by a 28 day timeline follow back.
  This outcome was corrected 3/2020 to accurately reflect the time frame from the original protocol. It was also moved to the secondary outcome measure section as was the original intent.
Alcohol-Related Negative Health Behaviors and Consequences: episodes of impaired drivin | 12 months post enrollment
  Self reported alcohol-related negative health behaviors and consequences based on the Brief Event Data survey (includes episodes of impaired driving, riding with an impaired driver, injuries, arrests, tardiness and days absent from work/school)
Alcohol-Related Negative Health Behaviors and Consequences: episodes riding with an impaired driver | 12 months post enrollment
  Self reported alcohol-related negative health behaviors and consequences based on the Brief Event Data survey (includes episodes of impaired driving, riding with an impaired driver, injuries, arrests, tardiness and days absent from work/school)
Alcohol-Related Negative Health Behaviors and Consequences: number of injuries | 12 months post enrollment
  Self reported alcohol-related negative health behaviors and consequences based on the Brief Event Data survey (includes episodes of impaired driving, riding with an impaired driver, injuries, arrests, tardiness and days absent from work/school)
Alcohol-Related Negative Health Behaviors and Consequences: number of arrests | 12 months post enrollment
  Self reported alcohol-related negative health behaviors and consequences based on the Brief Event Data survey (includes episodes of impaired driving, riding with an impaired driver, injuries, arrests, tardiness and days absent from work/school)
Alcohol-Related Negative Health Behaviors and Consequences: episodes of tardiness from work/school | 12 months post enrollment
  Self reported alcohol-related negative health behaviors and consequences based on the Brief Event Data survey (includes episodes of impaired driving, riding with an impaired driver, injuries, arrests, tardiness and days absent from work/school)
Alcohol-Related Negative Health Behaviors and Consequences: days absent from work/school | 12 months post enrollment
  Self reported alcohol-related negative health behaviors and consequences based on the Brief Event Data survey (includes episodes of impaired driving, riding with an impaired driver, injuries, arrests, tardiness and days absent from work/school)

OTHER OUTCOMES:
30 Day Treatment Engagement | 30 days post enrollment
  Engagement in alcohol treatment program based on Treatment Services Review at 30 day phone follow up

CONTACTS AND LOCATIONS:
Overall Officials: Federico Vaca, MD, MPH, Principal Investigator — Yale University
Locations (1):
- Bridgeport Hospital, Bridgeport, Connecticut, United States

REFERENCES:
- [Background] Vaca FE, Dziura J, Abujarad F, Pantalon MV, Hsiao A, Field CA, D'Onofrio G. Trial study design to test a bilingual digital health tool for alcohol use disorders among Latino emergency department patients. Contemp Clin Trials. 2020 Sep;96:106104. doi: 10.1016/j.cct.2020.106104. Epub 2020 Aug 7. PMID 32777381
- [Derived] Vaca FE, Dziura J, Abujarad F, Pantalon M, Hsiao A, Reynolds J, Maciejewski KR, Field CA, D'Onofrio G. Use of an Automated Bilingual Digital Health Tool to Reduce Unhealthy Alcohol Use Among Latino Emergency Department Patients: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2314848. doi: 10.1001/jamanetworkopen.2023.14848. PMID 37219901